CLINICAL TRIAL: NCT06294977
Title: Impact of COVID-19 Pandemic on Epilepsy Evaluations in the Pediatric Emergency Department
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Alberto Cappellari, Princpal investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: CRISI-COVID
Record Dates: First submitted 2024-03-04; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Epilepsy; Emergency Services, Hospital; COVID-19
MeSH Terms: conditions — Epilepsy; Emergencies; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Background. Seizures are a common cause of evaluation in the pediatric emergency department (ED). Several studies about the impact of COVID-19 pandemic on ED attendances report a considerable reduction in general pediatric care. The aim of our study was to evaluate the impact of COVID-19 on the admission to the pediatric ED for seizures.

Materials and methods. We performed a retrospective study to assess the rate of ED admission for seizures at the pediatric ED of the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico of Milan between January 2017 and December 2021, comparing the pre-pandemic (from January 2017 to February 2020) and pandemic periods (from March 2020 to December 2021).

ELIGIBILITY:
Inclusion Criteria:

* age: 1 months to 17 years
* sex: all
* with at least one access to the Pediatric ED of the hospital for seizures

Exclusion Criteria:

* children who received a diagnosis of seizure on admission in triage that was not confirmed at discharge (breath-holding spell, fainting…).

Ages: 1 Month to 17 Years | Sex: All
Age Groups: Child
Study Population: All children under the age of 18 years who had at least one access to the Pediatric ED of the hospital for seizures
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
During the study period, 1,091 patients with seizures were admitted to pediatric ED, 776 before the pandemic and 315 during the pandemic. In particular, the evaluation rates per month were 20.4 before the pandemic and 14.3 afterward | the pre-pandemic (from January 2017 to February 2020) and pandemic periods (from March 2020 to December 2021)

SECONDARY OUTCOMES:
Patients with a history of previous seizures showed a greater decrease in the monthly number of ED visits compared to those with a first seizure. An increased rate of unprovoked seizures and a decreased rate of provoked ones were observed in the pandemic | the pre-pandemic (from January 2017 to February 2020) and pandemic periods (from March 2020 to December 2021)

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Emergency Department Clinica de Marchi, Foundation IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy